CLINICAL TRIAL: NCT06191068
Title: A Prospective, Multi-centre, Observational Study to Evaluate Two Patient-reported Outcome Measures, in Boys With Moderate or Severe Hemophilia Receiving Long-term Hemostatic Prophylaxis
Brief Title: Canadian CHO-KLAT/H-FIT Study - Quality of Life of, and Burden of Caring for, Persons With Hemophilia
Status: Not yet recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Caroline Malcolmson, Principal Investigator, Staff Physician Division of Haematology/Oncology, The Hospital for Sick Children
Other Study IDs: 41238567
Record Dates: First submitted 2023-12-04; First posted 2024-01-05 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Hemophilia
Keywords: health-related quality of life; quality of life; burden of care
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary goal of this observational study is to determine if:

* health-related quality of life of boys with moderate/severe hemophilia A who are followed in Canadian pediatric hemophilia treatment centres is significantly different for boys receiving an intravenously administered factor replacement product compared to a subcutaneously administered non-factor replacement product, as measured at the 3 month time-point.
* Burden of caring for a boy with moderate/severe hemophilia A is significantly different for parents/caregivers of boys with moderate/severe hemophilia A receiving an intravenously administered factor replacement product compared to a subcutaneously administered non-factor replacement product, as measured at the 3 month time-point.

Persons with hemophilia and their caregivers will complete questionnaires at baseline, three months, six months, and one week after six months.

DETAILED DESCRIPTION:
Hemophilia A is an inherited bleeding disorder that affects 1/5000 live male births. Advances in hemophilia care through the development of recombinant standard and extended half-life (SHL and EHL, respectively) clotting factor concentrates (CFCs) have improved disease management; however, the burden of frequent administration of intravenous CFCs can contribute to negative physical and psychosocial outcomes in both the patient and their family. A new non-factor hemostatic agent (emicizumab) allows for subcutaneous injections, given on a schedule that ranges from once weekly to once monthly. Given the very high cost of preventive treatments ("prophylaxis") as advances in care of persons with hemophilia are made (e.g., EHL CFCs, emicizumab), it is imperative that the potential health outcome benefits of these treatments are assessed using relevant validated outcome measures. There are two patient-reported outcome measures (PROMs) that have been previously validated for use in boys with hemophilia using SHL or EHL CFCs and their parents: the Canadian Hemophilia Outcomes-Kids Life Assessment Tool version 3 (CHO-KLAT 3.0) assessing health-related quality of life for boys with hemophilia A ages 4-18, and the Hemophilia Family Impact Tool version 1.1 (H-FIT 1.1) assessing burden of caring for a child with hemophilia for parents of boys with hemophilia A ages 0-18 years. However, their use in the context of emicizumab has not been evaluated. As such, the primary aim of this study is to determine if health-related quality of life of boys with moderate/severe hemophilia A who are followed in Canadian pediatric HTCs is significantly different for boys receiving an intravenously administered factor replacement product compared to a subcutaneously administered non-factor replacement product, and to determine if burden of caring for a boy with moderate/severe hemophilia A is significantly different for parents/caregivers of boys with moderate/severe hemophilia A receiving an intravenously administered factor replacement product compared to a subcutaneously administered non-factor replacement product, as measured at the 3 month time-point.

Secondary aims include:

* To assess the validity of the CHO-KLAT 3.0/H-FIT 1.1 for use in the context of emicizumab.
* To determine the measurement properties of the CHO-KLAT 3.0 and the H-FIT 1.1, including the minimal clinical important difference, the test-retest reliability, and the standard error of measurement (SEM);
* To determine parents' satisfaction with emicizumab using the Emicizumab Preference (EmiPref) Survey;
* To translate the CHO-KLAT 3.0 and the H-FIT 1.1 to French (Canadian) and assess its validity.

Lastly, the investigators will explore the HRQoL and impact of hemophilia on boys with moderate/severe hemophilia A complicated by FVIII inhibitors, and their families. The investigators will also explore the use of the EmiPref and Parental Needs Scale for Rare Diseases (PNF-RD) in parents of boys with moderate/severe hemophilia to investigate their relationship with the disease-specific CHO-KLAT 3.0 and H-FIT 1.1, respectively.

The CHO-KLAT 3.0 is a validated, child-centric HRQoL measure for use in boys with hemophilia between the ages of 7-18 (self-report), and between the ages of 4-18 (parent-proxy report). The H-FIT 1.0 was developed to determine the impact of caring for a child with hemophilia from birth to 18 years on the family, and is especially relevant during the early years of diagnosis and initiation of primary prophylaxis. The H-FIT 1.1 was adapted following modifications during cognitive debriefing (ongoing). Additional tools that will be included in this study are the Pediatric Quality of Life-Core Module (PedsQL-Core), the Pediatric Quality of Life-Family Impact Module (PedsQL-FIM), the Parental Needs Scale for Rare Diseases (PNS-RD), and the Emicizumab Preference Survey (EmiPref). The PedsQL-Core is a validated, generic tool designed to measure the impact of having a chronic health condition on quality of life and will be used to determine construct validity of the hemophilia-specific CHO-KLAT 3.0. The PedsQL-FIM is a validated, generic tool designed to measure the impact of caring for a child with a chronic health condition on parents and the family and will be used to determine construct validity of the hemophilia-specific H-FIT 1.1. The PNS-RD is a measure of the supportive care needs of parents of children with rare diseases and its relationship with the H-FIT 1.1 will be explored. The EmiPref is an industry (Roche)-developed tool used to assess patients' treatment preference and will be used to examine patients' satisfaction with emicizumab compared to previous treatments. These measures will be translated into French (Canadian) prior to commencing data collection (Phase 1). Cognitive debriefing will be completed with boys (n=8) and parents (n=8) at one French-speaking site in Quebec to confirm the translated measures are clear and relevant. Questionnaires will be administered in a random order to account for order effects.

For all groups, reliability data will also be collected with a repeat administration of the CHO-KLAT 3.0 and H-FIT 1.1 within 7 days of the 6-month time point in study subjects in a non-bleeding state (by self-report on the study case report form) for a minimum of 2 weeks prior to the administration of the questionnaires, since reliability can only be determined if the health status of the participant has not changed between administrations. Only one parent/guardian will be requested to complete the questionnaires per family.

ELIGIBILITY:
Inclusion Criteria:

* Boys with moderate/severe hemophilia A, with or without FVIII inhibitors, age 7-18 years,

  * Group A: who have previously received prophylaxis with SHL or EHL CFCs at least once a week for the previous year who plan on switching or who have switched to emicizumab.
  * Group B: who are currently receiving prophylaxis at least once a week for the previous year with any form of treatment other than emicizumab who are not switching treatment regimens.
  * Group C: who have not been on long-term prophylaxis for the year prior to study commencement who begin prophylactic treatment with emicizumab (i.e., previously untreated patients or patients receiving treatment on demand).
  * Group D: boys with moderate/severe hemophilia A who have neutralizing alloantibodies to FVIII (FVIII inhibitors), defined as a level of ≥0.6 Bethesda Units (BU) using the Nijmegen modification of the Bethesda assay on two separate occasions within a 1-4 week period1, who are receiving a by-passing hemostatic agent such as a non-activated or activated plasma-derived, virus-inactivated prothrombin complex clotting factor concentrate (e.g., FEIBA), recombinant FVIIa (Niastase), or emicizumab. FVIII Inhibitors of <5 BU are considered low titer and those ≥5 BU are considered high titer.
* Parents/caregivers of boys with moderate/severe hemophilia A with or without FVIII inhibitors between the ages of 0-18 years.
* Moderate or severe hemophilia A, defined as FVIII activity level ≤5%.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.

Exclusion Criteria:

Candidates will be excluded from study entry if any of the following criteria exist at the time of screening, or at the time point specified in the individual criterion listed:

* Boys with mild hemophilia A, defined as a FVIII activity between 5-40%.
* Presence of significant comorbid diseases (e.g., HIV) as per the judgement of the clinical team.
* Inability to read, write, and/or understand English or French.
* Unable or unwilling to provide informed consent.

Ages: 1 Month to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will involve data collection on male patients 18 years of age or less with moderate or severe hemophilia A, on prophylaxis, with or without FVIII inhibitors, and their parents/guardians. Parents/guardians of boys <18 years with moderate or severe hemophilia A will also be included for the objectives that involve the H-FIT 1.1.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Differences in health-related quality of life between boys receiving an intravenously administered factor product compared to subcutaneous non-factor product. | 3 months
  The correlation of the CHO-KLAT scores for boys receiving an intravenously administered factor replacement product compared to a subcutaneously administered non-factor replacement product, as measured at the 3 month time-point. The Canadian Hemophilia Outcomes-Kids' Life Assessment Tool v3.0 has 41 questions. Items 1 to 28 are scored on a 5-point scale from 1 (Never) to 5 (Always). Items 29 to 41 are scored on the same 5-point scale, with an additional Not Applicable option. The tool is scored using a summary score of all items from 0 to 100, with 100 representing the best quality of life.
Differences in burden of caring for boys receiving an intravenously administered factor product compared to subcutaneous non-factor product. | 3 months
  The correlation of the H-FIT scores for parents/caregivers of boys receiving an intravenously administered factor replacement product compared to a subcutaneously administered non-factor replacement product, as measured at the 3 month time-point.
  The Hemophilia Family Impact Tool v1.1 has 25 questions scored on a 5-point scale from 1 (never) to 5 (always). The questionnaire is scored as a summary score of all items from 0 to 100, with 100 representing the lowest family burden.

SECONDARY OUTCOMES:
Validity of the CHO-KLAT and H-FIT | 6 months
  The secondary endpoints include the correlation of the CHO-KLAT 3.0 with the PedsQL-core module and the correlation of the H-FIT 1.1 with the PedsQL-FIM.
  The PedsQL 4.0-Generic Core Scale consists of 21 items covering 4 dimensions including physical functioning, emotional functioning, social functioning, and school functioning. Most items are scored on a 5-point scale from 0 (Never) to 4 (Almost always). The tool is scored using a summary score of all items from 0 to 100, with 100 representing the best quality of life. The PedsQL 2.0-Family Impact Module is a Parent report of family impact which is consisting of 36 items covering 8 dimensions. All items are score on a 5-point scale from 0 (Never) to 4 (Almost always). The tool is scored using a summary score of all items from 0 to 100, with 100 representing the best functioning.

IPD SHARING:
Plan to Share IPD: No